CLINICAL TRIAL: NCT03474237
Title: A Prospective Cohort Study for Patients With Adrenal Diseases
Status: Enrolling by invitation | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Hee Kim, Principal Investigator, Seoul National University Hospital
Other Study IDs: 1801-010-911
Record Dates: First submitted 2018-03-10; First posted 2018-03-22 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Adrenal Adenoma; Cushing Syndrome; Pheochromocytoma; Adrenal Incidentaloma; Adrenocortical Carcinoma; Primary Hyperaldosteronism
Keywords: algorithms; adrenal adenoma; cushing syndrome; pheochromocytoma; adrenal incidentaloma; adreocortical carcinoma; primary hyperaldosteronism
MeSH Terms: conditions — ACTH Syndrome, Ectopic; Cushing Syndrome; Pheochromocytoma; Adrenal incidentaloma; Adrenocortical Carcinoma; Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Non-functioning adrenal incidentaloma: patients who were diagnosed with non-functioning adrenal incidentaloma on computed tomography or magnetic resonance imaging
  Interventions: Other: Hormone study and Imaging study
- Pheochromocytoma: patients who were diagnosed with pheochromocytoma biochemically or histologically
  Interventions: Other: Hormone study and Imaging study
- Primary aldosteronism: patients who were diagnosed with primary aldosteronism by saline loading test
  Interventions: Other: Hormone study and Imaging study
- Adrenal cushing syndrome: patients who were diagnosed with adrenal cushing syndrome by dexamethasone suppression test and 24 urine free cortisol test.
  Interventions: Other: Hormone study and Imaging study
- Adrenocortical carcinoma: patients who were diagnosed with adrenocortical carcinoma by imaging study or histologic exam
  Interventions: Other: Hormone study and Imaging study

INTERVENTIONS:
Other: Hormone study and Imaging study — 1. Blood (basal hormone and follow up hormone study)
  2. Imaging examination including computed tomography scan or magnetic resonance imaging

SUMMARY:
The purpose of this study is to investigate the pathologic features, complications, and prognostic factors of functioning adrenal adenoma and suggest follow-up algorithms for adrenal incidentaloma.

DETAILED DESCRIPTION:
The investigators will recruit 150 patients annually for 10 years (adrenal incidentaloma 100 patients, pheochromocytoma 15 patients, primary aldosteronism 25 patients, adrenal cushing syndrome 10 patients, adrenocortical carcinoma 2 patients) and perform hormonal, biochemical, imaging exam according to each disease's clinical guidelines. Based on this, the investigators will identify pathologic features, complications, and prognostic factors of each disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults, male or female aged 19 years or older
* newly diagnosed with adrenal disease such as adrenal incidentaloma, pheochromocytoma, primary aldosteronism, adrenal cushing syndrome, adrenocortical carcinoma

Exclusion Criteria:

* previous or current history of adrenal diseases
* using oral or intravenous steroids
* history of major depressive disorder
* history of chronic alcoholics
* history of any cancer with suspicious adrenal metastasis
* those with acute illness (ex- patients with acute coronary syndrome within 4 weeks, acute febrile disease)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study population of this study is the patients who are newly diagnosed with adrenal disease such as adrenal incidentaloma, pheochromocytoma, primary aldosteronism, adrenal cushing syndrome, adrenocortical carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants in remission | Up to 10 years
  Remission rate

SECONDARY OUTCOMES:
Complication of adrenal disease | Up to 10 years
  all complications including deaths

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hee Kim, M.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No